CLINICAL TRIAL: NCT05316688
Title: Intraoperative Visualization of Oral Cavity Squamous Cell Carcinoma and High-Grade Dysplasia With Tozuleristide, a Fluorescent Tumor Marking Agent
Brief Title: A Fluorescent Tumor Marking Agent, Tozuleristide, for Imaging Oral Cavity Squamous Cell Cancer and High-Grade Oral Cavity Dysplasia During Surgery
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Blaze Bioscience Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RG1122110; NCI-2022-01734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020096 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Stage I Lip and Oral Cavity Cancer AJCC v8; Stage II Lip and Oral Cavity Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — tozuleristide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (tozuleristide, surgery, NIR imaging) (Experimental): Beginning 1 hour before surgery, patients receive tozuleristide intravenously (IV) over 1-5 minutes. Patients then surgical resection per standard of care and undergo near infrared (NIR) imaging with standard of care device.
  Interventions: Procedure: Near Infrared Imaging; Procedure: Therapeutic Conventional Surgery; Drug: Tozuleristide

INTERVENTIONS:
Procedure: Near Infrared Imaging — Undergo NIR imaging
  Other Names: Near-Infrared Imaging; NIR Imaging
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Drug: Tozuleristide — Given IV
  Other Names: BLZ-100

SUMMARY:
This phase I/II trial studies the side effects of tozuleristide in imaging oral cavity squamous cell cancer and high-grade oral cavity dysplasia during surgery. Tozuleristide is an imaging agent that specifically binds to tumor cells. When exposed to near-infrared light, tozuleristide causes tumor cells to fluoresce (light up), so that surgeons may better distinguish tumor cells from healthy cells during surgery.

DETAILED DESCRIPTION:
OUTLINE:

Beginning 1 hour before surgery, patients receive tozuleristide intravenously (IV) over 1-5 minutes. Patients then surgical resection per standard of care and undergo near infrared (NIR) imaging with standard of care device.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects age >= 18 years (yr)
* Subjects must have suspected or confirmed oral cavity dysplasia or cT1-4 squamous cell carcinoma for which surgical excision is deemed clinically indicated by the treating physician. Histology confirmation not required prior to surgery
* Able to provide written informed consent
* If of child-bearing potential, agree to the continued use of 2 reliable forms of contraception from study enrollment through 30 days after receiving the study product. Male subjects must agree to use 2 reliable methods of contraception simultaneously for 30 days after receiving the study product if their partner is of child-bearing potential
* Available for all study visits and able to comply with all study requirements

Exclusion Criteria:

* Known or suspected sensitivity to indocyanine green
* In the opinion of the treating physician, subject has received photosensitizing medication that could interfere or confound study results
* Any current medications with the potential to generate fluorescence or photochemical reaction
* Enrolled in any other ongoing study
* Currently lactating or breastfeeding
* Positive pregnancy test or planning to become pregnant within 30 days (d) of receiving tozuleristide
* Any current condition, including psychological and social situations which, in the opinion of the investigator, would impact adversely on the subject or the interpretation of the study data
* Creatinine clearance < 60 mL/min
* Aspartate aminotransferase (AST) > 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) > 1.5 x ULN
* Bilirubin > 1.5 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | 7-21 days after drug administration
  Adverse events will be summarized as the number and percentage of patients with each type of adverse event, per Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Number of subjects without tumor fluorescence after receiving tozuleristide | Up to 12 months
Sensitivity of tozuleristide fluorescence to detect tumor in tissue biopsies | Up to 12 months
  Will be estimated by a repeated measure logistic regression modeling the probability of positive tumor. The model includes an exchangeable working correlation structure to account for potential correlations of biopsies within subject for the tumor-positive tissue biopsies. A general estimating equation (GEE) method will be used to estimate the regression parameters.
Specificity of tozuleristide fluorescence to detect tumor in tissue biopsies | Up to 12 months
  Will be estimated by a repeated measure logistic regression modeling the probability of negative tumor. The model includes an exchangeable working correlation structure to account for potential correlations of biopsies within subject for the tumor-positive tissue biopsies. A GEE method will be used to estimate the regression parameters. The repeated measures logistic regression will model the probability of tumor-negative biopsies.
Positive predictive value of tozuleristide fluorescence to detect tumor in tissue biopsies | Up to 12 months
Negative predictive value of tozuleristide fluorescence to detect tumor in tissue biopsies | Up to 12 months
Achievement of negative margins in tozuleristide-guided oral cavity tumor excision | Up to 12 months
  To investigate the accuracy of tozuleristide fluorescent imaging in identifying tumor and achieving negative margins during excision of oral cavity squamous cell carcinoma and high-grade dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Marchiano, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No